CLINICAL TRIAL: NCT06606067
Title: Efficacy of Perioperative Duloxetine in Patients at High Risk for Developing Chronic Postsurgical Pain After Inguinal Hernia Repair: a Multicenter Randomized Controlled Trial.
Brief Title: Duloxetine to Prevent Chronic Postsurgical Pain After Inguinal Hernia Repair in Patients at High Risk
Acronym: GENDOLCAT3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Carlos III Health Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ICI21 / 00006; 2022-001354-29 (EudraCT Number)
Record Dates: First submitted 2024-09-04; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Chronic Post-surgical Pain
Keywords: Chronic post-surgical pain; Duloxetine; Prevention; Hernia repair
MeSH Terms: conditions — Pain, Postoperative | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Duloxetine Placebo
Who Masked: Participant, Investigator
Masking Description: Placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duloxetine (Experimental): Participants received Duloxetine 30 mg / 24 h 2 weeks before surgery and 1 week after surgery
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Participants received Placebo / 24 h 2 weeks before surgery and 1 week after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 30 mg daily 2 weeks before surgery and 1 week after surgery
  Arms: Duloxetine
Drug: Placebo — Placebo tablet daily
  Arms: Placebo

SUMMARY:
The clinical trial will be conducted in 14 Spanish hospitals. It is estimated, based on our previous studies, that 2855 patients scheduled for elective inguinal hernia surgery will have to be assessed to detect patients with ≥ 27% level of risk for Chronic Post-Surgical Pain (CPSP). These high-risk patients will be randomized to 2 treatment groups: one will receive duloxetine for 2 weeks prior to surgery and 1 week after surgery (intervention group) and the other the placebo (control group) during the same periods. The primary outcome will be a ≥ 50% decrease in the CPSP incidence in the intervention group compared to the placebo group, 4 months after surgery.

DETAILED DESCRIPTION:
Prospective, multicenter, double-blind randomized double-blind controlled trial. In the first phase the investigators use the Chronic Post-Surgical Pain (CPSP) risk model to select patients scheduled for inguinal hernia repair with a ≥27% level of risk for CPSP.

A total of 2855 patients will be screened in 14 Spanish hospitals (Hospital del Mar (Barcelona) / Hospital Germans Trias i Pujol (Badalona) / H Vall d'Hebrón (Barcelona) / Hospital de Bellvitge (Barcelona) / Hospital de Cruces (Bilbao) / Hospital 12 de Octubre (Madrid) / Hospital de Valme (Sevilla) / Hospital de Son Espases (Palma de Mallorca) / Hospital Son Llatzer (Palma de Mallorca) / Hospital General de Valladolid (Valladolid)/ Hospital General de Alicante (Alicante)/ Hospital Lluís Alcanyís de Xativa).

The high-risk patients will be randomized to 2 treatment groups to receive 30 mg/d of duloxetine for 2 weeks prior to surgery and 1 week after surgery (intervention group) or placebo (control group) during the same periods.

The primary outcome will be a decrease in the CPSP incidence at 4 months in the intervention group compared to the placebo group with an odds ratio of 0.44 as the effect size. The investigators estimate that it will be necessary to treat 294 participants (147 in each group). Participants that might have CPSP will be detected in follow-up telephone interviews approximately 3 months after surgery. Participants who report pain at that time will be scheduled for an appointment at their hospital's pain clinic to confirm the CPSP diagnosis by exhaustive physical examination and to assess pain intensity, characteristics, and degree of interference with daily living.

ELIGIBILITY:
Inclusion Criteria:

* Men resident in Spain who are scheduled for open inguinal hernia repair (inpatient or outpatient procedures).
* Risk of post-surgical pain chronification > 27% using the GENDOLCAT risk scale.

Exclusion Criteria:

* Age under 18 years
* Patients who in the recruiter's opinion have insufficient knowledge of Spanish to understand the trial
* Patients who are currently being treated with duloxetine
* Patents with known allergy to duloxetine
* Serious renal failure (creatinine clearance >30 ml/min)
* Patients requiring reoperation because of surgical complications
* Transplanted patients
* History of coronary artery disease, including previous myocardial infarction, angina, percutaneous transluminal coronary angioplasty
* History of congestive heart failure
* Currently taking a monoamine oxidase inhibitor or other medication with substantial interaction with duloxetine
* Antidepressant use within 4 weeks of study start
* Treatment with inhibitors of cytochrome P450 mixed-function oxidase system (CYP1A2): fluvoxamine, ciprofloxacin or enoxacin
* Uncontrolled hypertension
* Bipolar disorder
* History of seizures
* Elevated intraocular pressure or risk of acute glaucoma
* Treatment with selective serotonin reuptake inhibitors (SSRIs)
* Treatment with serotonin and noradrenaline reuptake inhibitors (SNRIs)
* Treatment with tricyclic antidepressants
* Treatment with triptans
* Treatment with antipsychotic drugs
* Treatment with dopamine antagonists
* Treatment with oral anticoagulant agents
* Treatment with Hypericum perforatum
* Major depression disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The score to establish risk for chronic post-surgical pain is validated only in men
Enrollment: 294 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of duloxetine versus placebo in reducing the incidence of Chronic Post-Surgical Pain (CPSP) at 4 months | 4 months after surgery
  The primary outcome will be a change in the Chronic Post-Surgical Pain (CPSP) incidence at 4 months in the intervention group compared to the placebo group with an odds ratio of 0.44 as the effect size. Criteria of CPSP: 1) The pain develops after a surgical procedure or increases in intensity after the surgical procedure, 2) the pain should be of at least 3 months' duration and significantly affected the quality of life, 3) the pain is either a continuation of acute post-surgery pain or develops after an asymtomatic period, 4) the pain is either localized to the surgical field, projected to the innervation territory of a nerve situated in the surgical field, or referred to a dermatome, 5) other causes of the pain should be excluded: infection or continuing malignancy in cancer surgery.

SECONDARY OUTCOMES:
Characteristics of Chronic Post-Surgical Pain (CPSP) | 4 months after surgery
  Compare the characteristics of Chronic Post-Surgical Pain (CPSP) in the intervention and control groups with neuropathic pain questionnaire (Douleur Neuropathique 4 (DN4 spanish version).
Intensity of Pain | 4 months after surgery
  Compare the intensity characteristics of Chronic Post-Surgical Pain (CPSP) with Brief Pain Inventory-Short Form (BPI-SF).
Quality of life in patients with Chronic Post-Surgical Pain (CPSP) | 4 months after surgery
  Compare the quality of life in the intervention and control groups with the SF-12 questionnaire (validated Spanish version 2)
Adverse effects of perioperative duloxetine comparing with placebo | 2 weeks before surgery and 1 week after surgery
  Comparing the rates of adverse effects of perioperative duloxetine and placebo for the primary prevention of Chronic Post-Surgical Pain (CPSP).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Montes, PhD, Principal Investigator — Hospital del Mar Research Institute
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No